CLINICAL TRIAL: NCT06681415
Title: A Randomized Controlled Trial on the Efficacy of 20% Human Albumin in Reducing Pleural Effusion After Cardiopulmonary Bypass
Brief Title: Efficacy of 20% Human Albumin in Reducing Pleural Effusion After Cardiopulmonary Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Collaborators: Riga Stradins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PaulsStradins
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Pleural Effusions Post Coronary Artery Bypass Graft; Hypoxia; Hypoalbuminemia
Keywords: Pleural effusion following cardiopulmonary bypass
MeSH Terms: conditions — Hypoxia; Hypoalbuminemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin group (Experimental): The standard CPB priming volume of 1050 ml, comprising isochloremic solution Deltajonin® and 250 ml of 15% Mannitol, was used. The study group replaced 100 ml of Deltajonin® solution with 100 ml of 20% human albumin.
  Interventions: Drug: Adding 100ml of 20% human albumin to cardiopulmonary bypass priming solution
- No-albumin group (No Intervention): The standard CPB priming volume of 1050 ml, comprising isochloremic solution Deltajonin® and 250 ml of 15% Mannitol

INTERVENTIONS:
Drug: Adding 100ml of 20% human albumin to cardiopulmonary bypass priming solution — Adding albumin to the priming solution can help reduce hemodilution and consequent extracardiac complications by maintaining colloid oncotic pressure. Albumin helps counteract the intravascular fluid shift to the extravascular space and reduces the risk of complications associated with fluid imbalance.
  Postoperative pulmonary complications following CPB can significantly impact postoperative outcomes. Patients developing PPC have prolonged mechanical ventilation, extended hospitalisation, longer ICU stays, and elevated postoperative mortality. One of the most common PPCs following CPB is pleural effusion.
  Our primary objective was to evaluate the effectiveness of adding 100 ml of 20% human albumin to the CPB priming solution compared to standard priming, with a specific focus on its potential role in reducing the occurrence of pleural effusion.
  Arms: Albumin group

SUMMARY:
Human albumin is a widely used additive in cardiopulmonary bypass all around the world, but its effect on various outcomes has been debated. The goal of this observational study is to compare the effect of 100 ml 20% human albumin addition to cardiopulmonary bypass on pleural effusion development after open heart surgery.

The main question it aims to answer is:

• Does albumin, in addition to cardiopulmonary bypass, reduce pleural effusion development after open heart surgery? Patients will go under elective open heart surgery. Investigators will compare pleural effusion volume on the first day after surgery between patients who received albumin and those who didn't.

DETAILED DESCRIPTION:
This study constituted a prospective single-center randomized controlled trial conducted at the Center of Cardiac Surgery within Pauls Stradins Clinical University Hospital, Riga, Latvia. The study received approval from the State Agency of Medicines of the Republic of Latvia on September 20, 2021 for a drug usage observation study and the medical ethics committee of Pauls Stradins Clinical University Hospital (Chairperson Prof P. Stradins) under reference number 260821-11L, dated August 26, 2021. All participants provided written informed consent before enrolment.All participants provided written informed consent before enrolment.

The study targeted 70 individuals scheduled for elective open-heart surgeries, encompassing procedures such as ascending aorta surgery, coronary artery bypass grafting, and heart valve replacement or repair, either independently or in combination, without the use of hypothermic circulatory arrest. Investigators did not include patients with a history of reduced left ventricular ejection fraction (EF < 50%), chronic kidney disease, chronic lung disease, pre-existing anemia, and pathological chest X-ray findings before surgery. Random allocation into the two groups-those receiving an additional 100 ml of 20% human albumin and those receiving standard CPB priming solution-was done in a 1:1 ratio.

Interventions The standard CPB priming volume of 1050 ml, comprising isochloremic solution Deltajonin® and 250 ml of 15% Mannitol, was used. The study group replaced 100 ml of Deltajonin® solution with 100 ml of 20% human albumin. Investigators used cold crystalloid cardioplegia in all cases. Patients were mechanically ventilated according to the local protocol using FiO2 - 0.6, 6 ml/kg tidal volume, and PEEP was set at five mmHg. After extubation, oxygen was administered via a non-rebreathing face mask at a flow rate of 10 l/min. Blood gas analysis (pO2, pCO2, FiO2/O2 ratio, A - a gradients, Lactate) was conducted following the local protocol. Serum albumin levels were measured preoperatively, 6 and 12 hours post-operation. Normal albumin was defined as ≥35 g/L, mild 30-35 g/L, moderate 25-30 g/L and severe hypoalbuminemia as <25 g/L. Colloid oncotic pressure (COP) was calculated using the formula by J C Hoefs: COP = A (1.058 G + 0.163 A + 3.11).

Thorax CT scans were performed on all patients on the first postoperative day, with subsequent image analysis conducted by a single radiologist. The radiologist measured pleural effusion size (cm), and investigators calculated effusion volume (ml) using the formula Volume = 0.365 × b^3 - 4.529 × b^2 + 159.723 × b - 88.377 by Hazlinger et al. Where b is the maximum effusion depth measured in the axial (transverse) imaging plane. If patients were hemodynamically unstable with ST-segment abnormalities, investigators refused their transportation to a CT scan.

The primary outcomes were the effect of albumin addition on serum albumin level in the early postoperative period and the development of pleural effusion.

The secondary outcome measure was the effect of albumin addition on respiratory function, measured by blood gas analysis, in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals scheduled for elective open-heart surgeries, encompassing procedures such as ascending aorta surgery, coronary artery bypass grafting, and heart valve replacement or repair, either independently or in combination, without the use of hypothermic circulatory arrest.

Exclusion Criteria:

* reduced left ventricular ejection fraction (EF < 50%),
* chronic kidney disease,
* chronic lung disease,
* pre-existing anemia,
* pathological chest X-ray findings before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Pleural effusion (centimetres) in thoracic CT images and calculated in millilitres. | Thorax CT scans were performed on all patients on the first postoperative day.
  Thorax CT scans were performed on all patients on the first postoperative day, with subsequent image analysis conducted by a single radiologist. The radiologist measured pleural effusion size (cm).
Pleural effusion in thoracic CT images and calculated in millilitres. | Thorax CT scans were performed on all patients on the first postoperative day.
  Thorax CT scans were performed on all patients on the first postoperative day, with subsequent image analysis conducted by a single radiologist. The investigators calculated effusion volume (ml).

CONTACTS AND LOCATIONS:
Overall Officials: Eva Strike, MD, PhD, Study Director — Head of the cardiac anesthesiology and ICU department
Locations (1):
- Pauls Stradiņš Clinical University Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No